CLINICAL TRIAL: NCT06875141
Title: DM199 for Pregnancy Complications
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This entry was unauthorized and has been withdrawn.
Sponsor: DiaMedica Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PACTR202404895013782
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — DM199

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1 (Experimental): Part 1
  Interventions: Biological: DM199

INTERVENTIONS:
Biological: DM199 — DM199 is a synthetic form of rhKLK1

SUMMARY:
This entry was submitted in error by DiaMedica Therapeutics, Inc. and was not authorized by any of the trial Investigators or study sponsor (Stellenbosch University).

The clinical trial, DM199 for Pregnancy Complications, was prospectively registered with the Pan African Clinical Trials Registry (PACTR202404895013782), in accordance with ICMJE and WHO requirements. This listing serves as the primary and authoritative registration record for this investigator-initiated study.

ELIGIBILITY:
Please refer to the Pan African Clinical Trials Registry (PACTR202404895013782).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment adverse events | Until 6 weeks after the due date

IPD SHARING:
Plan to Share IPD: No